CLINICAL TRIAL: NCT06823011
Title: Effects of Banned Substances on Some Metabolic Functions in Male Amateur Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, LEVENT CEYLAN, associate professor, Hitit University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Hitit Üniversitesi
Record Dates: First submitted 2024-12-20; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Effects of Banned Substances
Keywords: Banned Substances; doping; anabolic steroid
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: group doing weight training and using banned substances
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group using banned substances (Other): group doing weight training and using banned substances
  Interventions: Diagnostic Test: blood collection
- group not using banned substances (Other): a group that does weight training but does not use banned substances
  Interventions: Diagnostic Test: blood collection

INTERVENTIONS:
Diagnostic Test: blood collection — Blood was collected from the study group and the control group at 10 am in the morning on an empty stomach.

SUMMARY:
The aim of this study was to investigate the effects of banned substances on some metabolic functions in male athletes in order to raise awareness among individuals who use these substances by highlighting the potential harms of using banned substances to draw attention to the issue and raise awareness. 2) Methods: The study is a randomised cross-sectional study. The study included 20 male amateur athletes who had actively practised bodybuilding, arm wrestling, powerlifting and weightlifting in the last 5 years and had not participated in competitions. The study group consisted of 10 adult male amateur athletes who had used banned substances at least once a year in the past 5 years, while 10 male amateur athletes who had not used banned substances with similar qualifications formed the control group. Participants were included in the study on a voluntary basis. Participants' age, sports age, height, weight and BMI variables were selected and parameters related to liver, kidney, hormone and lipid profiles were determined. The Shapiro-Wilk test was used to test the normality of the values obtained from the data. The independent t-test was used for the data showing a normal distribution and the Mann Whitney U- test was used for the data not showing a normal distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Amateur athlete who has been actively involved in bodybuilding, arm wrestling, powerlifting and weightlifting for the last 5 years
2. Adult male amateur athletes who use banned substances in at least 1 period each year

Exclusion Criteria:

1. with chronic illness
2. receiving continuous medication
3. heavy labor
4. who has recently had an infection
5. amateur athletes who performed heavy exercise in the last 72 hours

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 20 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
body mass index BMI in Male Athletes | 6 months, 1 year
  Height, body weight (BW), body mass index [BMI= BW (kg) / (height, m)2] were determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit Üniversity gym, Sivas, Si̇vas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are available on request from the corresponding author. The data are not publicly available due to restrictions related to ongoing work for further publications